CLINICAL TRIAL: NCT03153215
Title: Evaluation of Addition of Sildenafil Citrate for Treatment of Severe Intrauterine Growth Restriction
Brief Title: Sildenafil in Sever Intrauterine Growth Retardation
Acronym: IUGR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Nesreen Abdel Fattah Abdullah Shehata, Assistant Professor of Obstetrics and Gynecology, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Beni-Suef 12
Record Dates: First submitted 2017-05-05; First posted 2017-05-15 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Intra-Uterine Growth Retardation
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: A total of 46 patients with severe early onset intrauterine growth retardation will be enrolled in a randomized placebo control controlled study .
  Patients will randomly be allocated to two groups with 23 patients in each group
Who Masked: Participant, Investigator
Masking Description: Patients will randomly be allocated to two groups with 23 patients in each group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): women with severe IUGR
  Interventions: Other: treatment
- Control group (Active Comparator): women with severe IUGR
  Interventions: Other: Placebo

INTERVENTIONS:
Other: treatment — We will offer Sildenafil citrate (20 mg per os three times daily until delivery) as innovative therapy to 23 women with severe IUGR ('Sildenafil-treated') in addition to fish oil and zinc supplementation.
  Arms: Intervention group
Other: Placebo — Placebo tablets similar to Sildenafil will be given to control group in addition to fish oil and zinc supplementation.
  Arms: Control group

SUMMARY:
Severe fetal growth restriction (FGR) complicates approximately 0.4% of pregnancies and severely increases the risk of perinatal morbidity and mortality.Sildenafil citrate may offer a potential therapeutic strategy to improve uteroplacental blood flow in IUGR pregnancies.

DETAILED DESCRIPTION:
The aim of our study is to evaluate the effect of sildenafil citrate therapy on severe early and late onset intrauterine growth retardation.A total of 46 patients with severe early onset intrauterine growth retardation will be enrolled in a prospective case control study .

Patients will randomly be allocated to two groups with 23 patients in each group.Sildenafil citrate therapy may increase the likelihood of increased growth velocity [measured by abdominal circumference (AC) (ultrasound)] for fetuses of pregnancies complicated by severe early-onset IUGR .Sildenafil is a potent and selective inhibitor of cGMP-specific phosphodiesterase type 5 (PDE5), which is responsible for degradation of cGMP which results in increased levels of cGMP, leading to smooth muscle relaxation. Placental disease, consequent on deficient uteroplacental blood flow, includes FGR, pre-eclampsia, and placental abruption and has been implicated in more than 50% of iatrogenic premature births .For this reason, the problem of severe FGR forms a substantial portion of the population that tertiary care centres care.

ELIGIBILITY:
Inclusion Criteria:

• pregnancy complicated by severe IUGR [abdominal circumference (AC)< 5th percentile] the gestational age <25 weeks or an estimate of the fetal weight was <600 gm (excluding known fetal anomaly/syndrome and/or planned termination) ( von Dadelszen.et al;2011).

Exclusion Criteria:

* known aneuploid anomaly, syndrome congenital infection.
* If there is a plan to terminate the pregnancy.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2017-05-06 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Umbilical artery Pulsatility index | between 24 gestational weeks until 36 weeks
  Change in umbilical artery pulsatility index after medication
Middle cerebral artery Pulsatility index | between 24 gestational weeks until 36 weeks
  Change in middle cerebral artery pulsatility index after medication
fetal abdominal circumference growth velocity | between 24 gestational weeks until 36 weeks
  proportion of women in each group for whom fetal AC growth velocity will change post randomization.

SECONDARY OUTCOMES:
Rate of drug side effects | between 24 and 36 gestational weeks
  Women in the Sildenafil-treated group will be also monitored for adverse side-effects, such as flushing, lightheadedness and visual disturbance
Birth weight | between 24 and 36 gestational weeks
  weight of neonate at birth in grams

CONTACTS AND LOCATIONS:
Overall Officials: Nesreen A Shehata, MD, Principal Investigator — Beni-Suef University
Locations (1):
- Beni-Suef University, Cairo, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ananth CV, Vintzileos AM. Maternal-fetal conditions necessitating a medical intervention resulting in preterm birth. Am J Obstet Gynecol. 2006 Dec;195(6):1557-63. doi: 10.1016/j.ajog.2006.05.021. Epub 2006 Oct 2. PMID 17014813
- [Background] Lausman A, Kingdom J; MATERNAL FETAL MEDICINE COMMITTEE. Intrauterine growth restriction: screening, diagnosis, and management. J Obstet Gynaecol Can. 2013 Aug;35(8):741-748. doi: 10.1016/S1701-2163(15)30865-3. English, French. PMID 24007710
- [Background] Lee MJ, Conner EL, Charafeddine L, Woods JR Jr, Del Priore G. A critical birth weight and other determinants of survival for infants with severe intrauterine growth restriction. Ann N Y Acad Sci. 2001 Sep;943:326-39. doi: 10.1111/j.1749-6632.2001.tb03813.x. PMID 11594552